CLINICAL TRIAL: NCT03211455
Title: Effect of Continuous Intravenous Lidocaine on Early Rehabilitation in Bariatric Surgery. A Randomized Double Blind Controlled Study
Brief Title: Intravenous Lidocaine in Bariatric Surgery.
Acronym: XYLOBAR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-014
Record Dates: First submitted 2017-05-31; First posted 2017-07-07 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-05

CONDITIONS: Morbid Obesity; Bariatric Surgery Candidate
Keywords: bariatric surgery; rehabilitation; lidocaine
MeSH Terms: conditions — Obesity, Morbid | interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): intravenous isotonic saline administration : bolus of 0.075 ml/kg (adjusted body weight) at induction of anesthesia followed by a continuous infusion (0.1 ml/kg/h, adjusted body weight) until the end of surgery decrease to 0.05 ml/kg (adjusted body weight) during 60 min in post anesthesia care unit.
  Speed of infusion were calculated to be equivalent to that of lidocaine speed of injection.
  Interventions: Drug: isotonic saline
- Lidocaine (Experimental): Intravenous Lidocaine (20mg/ml) : bolus of 1.5 mg/kg (adjusted body weight) at induction of anesthesia followed by a continuous infusion (2.0 mg/kg/h, adjusted body weight) until the end of surgery decrease to 1.0 mg/kg (adjusted body weight) during 60 min in post anesthesia care unit.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — intravenous lidocaine versus placebo
  Arms: Lidocaine
Drug: isotonic saline — intravenous isotonic saline
  Other Names: saline
  Arms: Control

SUMMARY:
Although peroperative intravenous lidocaine has been shown to be useful in early recovery after colorectal surgery, its beneficial effect on the specific population of obese patients scheduled for bariatric surgery remained unknown.

Investigators hypothesized that peroperative intravenous lidocaine could decrease postoperative opioid consumption and improve postoperative recovery

DETAILED DESCRIPTION:
This is a prospective, double-blind, placebo-controlled, monocentric study. We plan to recruit 180 obese adult patients scheduled for bariatric surgery in a the french university hospital of Caen.

Exclusion: contra-indications for any aminoamide local anesthetic (allergy, severe hepatic disease) and for intravenous lidocaine (porphyria, atrioventricular conduction disturbances, uncontrolled seizure disease), long term opioid consumption, need for a post-operative follow-up in an intensive care unit, combined surgical procedure excepting cholecystectomy, pregnancy.

Patients will be randomly allocated to receive either a saline placebo or lidocaine continuous infusions during surgery. Morphinic consumption will be assessed from the end of the procedure until the third day after surgery. Secondary criteria will concern post-operative recovery, pain and postoperative nausea and vomiting, other medical and surgical complications, and toxicity. Plasma lidocaine concentrations will be measured in patients who had received lidocaine in order to determine the safety and efficiency of our infusion protocol.

Our analysis will be a superiority one, alpha risk is 5% and beta risk is 20%, in intention to treat, with no intermediate analysis.

ELIGIBILITY:
Inclusion Criteria:

* scheduled bariatric surgery

Exclusion Criteria:

* any contra-indication for lidocaine administration
* pregnancy
* ASA class 4
* psychiatric disorder
* chronic opioid consumption

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
oxycodone consumption | three days following surgery
  total postoperative (until day 3) oxycodone consumption (mg)

SECONDARY OUTCOMES:
lidocaine plasma concentration | during post anesthesia care unit stay (1 day)
  lidocaine plasma concentration measured at the end of infusion
hospital discharge check list | three days following surgery
  recovery (in days) which enable discharge from hospital
postoperative pain | three days following surgery
  postoperative pain intensity (visual analogue scale)
nausea and vomiting | three days following surgery
  proportion of patients with and without postoperative nausea and vomiting
intestinal transit recovery | three days following surgery
  duration (in days) of postoperative intestinal palsy
hospital length of stay | through hospital discharge (an average of 1 week)
  hospital length of stay

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Caen, Caen, France

IPD SHARING:
Plan to Share IPD: No